CLINICAL TRIAL: NCT03562533
Title: Comparison of Real-World Effectiveness of Pegylated Liposomal Doxorubicin Versus Paclitaxel in Platinum- Sensitive Recurrent Ovarian Cancer
Brief Title: Real-World Effectiveness of PLD in Platinum- Sensitive Recurrent Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); National Cancer Center, Korea (Other Government); Asan Medical Center (Other); The Catholic University of Korea (Other); Samsung Medical Center (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Ajou University (Other); Severance Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KUH1040075
Record Dates: First submitted 2018-05-23; First posted 2018-06-19 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin; 1-dodecylpyridoxal; Carboplatin; CP protocol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pegylated liposomal doxorubicin + carboplatin: carboplatin area under the curve [AUC] 5 plus pegylated liposomal doxorubicin (PLD) 30 mg/m2 every 4 weeks
  Interventions: Drug: pegylated liposomal doxorubicin (PLD) + carboplatin (CD)
- paclitaxel + carboplatin: carboplatin AUC 5 plus paclitaxel 175 mg/m2 every 3 weeks
  Interventions: Drug: carboplatin + paclitaxel (CP)

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin (PLD) + carboplatin (CD) — carboplatin AUC 5 plus paclitaxel 175 mg/m2 every 3 weeks for at least 6 cycles
  Groups: pegylated liposomal doxorubicin + carboplatin
Drug: carboplatin + paclitaxel (CP) — carboplatin AUC 5 plus paclitaxel 175 mg/m2 every 3 weeks for at least 6 cycles
  Groups: paclitaxel + carboplatin

SUMMARY:
This retrospective multicenter study aimed to evaluate the effectiveness of pegylated liposomal doxorubicin (PLD) with carboplatin (CD) compared with carboplatin and paclitaxel (CP) in patients who had disease progression longer than 6 months after first-line platinum+taxane chemotherapy for ovarian cancer in real world clinical practice.

DETAILED DESCRIPTION:
Worldwide, ovarian cancer is the sixth most common cancer and the seventh most common cause of cancer deaths in women. At the time of presentation, approximately 70% of women have advanced disease. Despite standard treatment of initial debulking surgery followed by chemotherapy in advanced ovarian cancer, most patients relapse after achieving a complete clinical response. Disease that responds to first-line therapy but relapses after 6 months after completion of initial platinum-based therapy is considered platinum sensitive (PS). Chemotherapy re-treatment is an important aspect in the overall management of patients with PS relapsed or recurrent ovarian cancer (ROC). Platinum is a backbone of treatment, and carboplatin and paclitaxel (CP) have emerged as standard in the first-line setting and been rechallenged in patients with platinum-sensitive ROC. A pooled analysis of three phase III trials from the AGO-OVAR and International Collaborative Ovarian Neoplasm collaborators demonstrated significant improvements in progression-free survival (PFS; hazard ratio [HR], 0.76; 95% confidence interval [CI], 0.66 to 0.89; P = .0004) and overall survival (OS; HR, 0.82; 95% CI, 0.69 to 0.97; P = .02) in patients with PS ROC treated with platinum-paclitaxel versus conventional platinum based therapies, mainly carboplatin monotherapy.

However, rechallenge with CP has been limited by the risk of cumulative peripheral neuropathy. In addition, grade 2 alopecia (complete hair loss), another ill-tolerated adverse effect for patients facing the distress of relapse, occurs in more than 80% of patients. In order to improve the patient's tolerance on the treatment in this setting, other carboplatin-based combinations, such as gemcitabine and carboplatin, have been explored. This combination significantly improved PFS versus carboplatin alone in phase III trial (HR, 0.72; 95%CI, 0.58 to 0.90; P= .0031). however, OS was not significantly improved (HR, 0.96; 95% CI, 0.75 to 1.23; P = .735); the trial was not powered to detect a survival difference. Grade 3 to 4 hematologic toxicities were significantly more frequent in the combination arm. Thus, a need for other carboplatin combinations remains in PS ROC.

Pegylated liposomal doxorubicin (PLD) is an active drug in ROC as the efficacy has been demonstrated in CALYPSO trial.

CAYPSO is a large randomized phase III showing the noninferiority of the combination of pegylated liposomal doxorubicin (PLD) with carboplatin (CD) compared with CP in patients with PS ROC. In this trial, PFS for the CD arm was statistically superior to the CP arm (hazard ratio, 0.821; 95% CI, 0.72 to 0.94; P = .005); median PFS was 11.3 versus 9.4 months, respectively. Overall severe nonhematologic toxicity (36.8% v 28.4%; P = .01) leading to early discontinuation (15% v 6%; P = .001) occurred more frequently in the CP arm. More frequent grade 2 or greater alopecia (83.6% v 7%), hypersensitivity reactions (18.8% v 5.6%), and sensory neuropathy (26.9% v 4.9%) were observed in the CP arm; more hand-foot syndrome (grade 2 to 3, 12.0% v 2.2%), nausea (35.2% v 24.2%), and mucositis (grade 2-3, 13.9% v 7%) in the CD arm.

Moreover, recent subgroup analysis of CALYPSO trial had reported that CD had a more favorable risk-benefit profile than CP in patients with partially platinum-sensitive ROC (patients with a treatment-free interval of >6 and ≤12 months). The hazard ratio for PFS was 0.73 (95% CI: 0.58-0.90; P = 0.004 for superiority) in favor of CD.

On the basis of the results of CALYPSO trial, Korea Food & Drug Administration (KFDA) has approved and reimbursed the use of PLD in patients with PS ROC since August 2014. From then, approximately 700 patients with PS ROC have been treated with PLD in Korea.

The majority of patients enrolled in CALYPSO have 1 prior treatment, however, CD has been used in diverse setting of ROC in Korea. Therefore, the effectiveness and safety of the PLD combination should be still evaluated in the real clinical practice in Korea. To fulfill the gap of knowledge between clinical trials and actual clinical practice, we perform a multicenter, retrospective, observational study of CD therapy in the second line setting of PS ROC.

ELIGIBILITY:
Inclusion Criteria:

* Previous taxane therapy was required.
* Recurred >6 months after surgery and first-line platinum-based chemotherapy regimen
* Patients with measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) or CA-125 assessable disease according to Gynecologic Cancer InterGroup (GCIG) criteria or histologic proven diagnosis
* Eastern Cooperative Oncology Group performance status of ≤ 2

Exclusion Criteria:

* Had ovarian tumors of low malignant potential (borderline tumors); nonepithelial or mixed epithelial/nonepithelial tumors (eg, mixed Mullerian tumors)
* Had received prior radiotherapy; or, had a previous diagnosis of malignancy within the past 5 years.
* Had bowel obstruction or presence of symptomatic brain metastases
* Patients with severe active infection
* Had history of severe hypersensitivity reactions to compounds chemically related to study products.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: A histologically confirmed diagnosis of epithelial ovarian, tubal, and primary peritoneal cancer, and recurred >6 months after first-line platinum-based chemotherapy regimen
Sampling Method: Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 36 months
  OS was defined as the time from randomization to death of any cause. The OS data for participants for whom no death was captured in the clinical database were censored at the last time they were known to be alive.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 3years
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the investigators according to the RECIST criteria.
Incidence of Treatment-Related Adverse Events | 36 months
  Safety and tolerability will be assessed in deaths, laboratory data, and vital signs. Number of participants with treatment-related adverse events as assessed by CTCAE version 4.0.
Response rate | 36 months
  Best Overall Confirmed Objective Response of Complete Response (CR) or Partial Response (PR) by Modified RECIST until progression reported. Objective Response was determined by the investigator using modified RECIST criteria, Version 1.0. An objective response was a complete or partial overall confirmed response as determined by investigators. CR defined as complete disappearance of all target and non-target lesions and no new lesions. PR defined as greater than or equal to (≥) 30 percent (%) decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyuk Shim, MD, Principal Investigator — Konkuk University Hospital
Locations (1):
- Konkuk University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SJ, Kim J, Kim HS, Lee JW, Chang HK, Lee KH, Kim DY, Kim S, Chang SJ, Han SS, Park SY, Shim SH. Real world effectiveness and safety of pegylated liposomal doxorubicin in platinum-sensitive recurrent ovarian, fallopian, or primary peritoneal cancer: a Korean multicenter retrospective cohort study. J Gynecol Oncol. 2020 Mar;31(2):e15. doi: 10.3802/jgo.2020.31.e15. Epub 2019 Sep 10. PMID 31912673